CLINICAL TRIAL: NCT01132885
Title: Defining the Brain Phenotype of Children With 7q11.23 Copy Number Variation, Including Williams Syndrome and 7q11.23 Duplication Syndrome
Brief Title: Defining the Brain Phenotype of Children With Williams Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100112; 10-M-0112
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-05-14

CONDITIONS: Williams Syndrome; Duplication
Keywords: MRI; Developmental; Genetic abnormalities in chromosome 7q11.23.; Duplication; Brain; Natural History; Williams Syndrome; Children; Healthy Volunteer; HV
MeSH Terms: conditions — Williams Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Adults with WS or genetic abnormalities: Adults with Williams syndrome or genetic abnormalities in chromosome 7q11.23
- Children with WS or genetic abnormalities: children ages 5-17 with Williams Syndrome or genetic abnormalities in chromosome 7q11.23
- Parents: Parents of children with 7q11.23 CNV will undergo blood draws
- Unaffected Siblings: Siblings of children with 7q11.23 CNV
- Unrelated children: Typically developing children ages ages 5-17

SUMMARY:
Background:

- Little is known about how the brain changes during childhood and adolescence, how genes affect this process, or how the brains of people with 7q11.23 genetic variation change during this period. Researchers are interested in using magnetic resonance imaging to study how the brain changes in healthy children and children with 7q11.23 genetic variation, including Williams syndrome and 7q11.23 duplication syndrome.

Objectives:

- To study developmental changes in the brains of healthy children and children who have been diagnosed with Williams syndrome,7q11.23 duplication syndrome, or other 7q11.23 genetic variation.

Eligibility:

* Healthy children and adolescents between 5 and 17 years of age.
* Children and adolescents between 5 and 17 years of age who have been diagnosed with Williams syndrome, 7q11.23 duplication syndrome, or have other 7q11.23 genetic variation.

Design:

* Participants will have a brief physical examination and tests of memory, attention, concentration, and thinking. Parents will be asked about their child s personality, behavior characteristics, and social interaction and communication skills.
* Both participants and their parents may be asked to complete additional questionnaires or take various tests as required for the study.
* Participants will have approximately 10 hours of magnetic resonance imaging (MRI) scanning, usually over 4 to 5 days, within a one month period. Some of these tests will require the participants to do specific tasks while inside the MRI scanner.
* Participants will be asked to return to the National Institutes of Health clinical center to repeat these procedures every 2 years thereafter until age 18.

DETAILED DESCRIPTION:
Williams syndrome is a rare disorder caused by hemizygous microdeletion of approximately 1.6 megabases on chromosomal band 7q11.23, typically by spontaneous mutation. The disorder is characterized by a collection of unique neuropsychiatric manifestations, including marked visuospatial construction deficits and hypersociability. Because the genes involved in WS are known, the study of neural mechanisms in WS affords a privileged setting for investigating genetic influences on complex brain functions in a bottom-up way.

Previous neuroimaging studies of adults with Williams syndrome resulted in a clear delineation of the Williams syndrome brain phenotype. Underlying the syndrome s cognitive hallmark, visuospatial construction impairment, is a neurostructural anomaly (decreased gray matter volume) and adjacent abnormal neural function in the parietal sulcus region of the dorsal visual processing stream. Subtle structural hippocampal alterations, along with abnormalities in regional cerebral blood flow, neurofunctional activation, and N-acetyl aspartate concentration also contribute to the visuospatial phenotype. Underlying the syndrome s social cognition features are structural and functional abnormalities in the orbitofrontal cortex, an important affect and social regulatory region that participates in a fronto-amygdala regulatory network found to be dysfunctional in Williams syndrome.

The findings in adult Williams syndrome patients have created a paradigm for identifying brain phenotypes linked to specific genes and for guiding research aimed at understanding the mechanism by which gene effects are translated in the brain to clinical phenomena. However, it is clear that the cognitive and behavioral disturbances in Williams syndrome emerge over the course of childhood and adolescence from a complex interplay of altered neural systems, which must be studied from a developmental and translational perspective. To meet this imperative, we propose a cross-sectional and longitudinal neuroimaging study of children with Williams syndrome to track the emergence and modification of the altered neural circuitry observed in the adult population. With non-invasive multimodal magnetic resonance imaging including structural MRI, functional MRI (fMRI), and diffusion tensor MRI-we propose to target those neural systems associated with key clinical features (e.g. visuospatial construction impairment and abnormal social cognition). We will employ experimental methods previously successful in assessing cognitive and emotional processing in the adult population. For neurofunctional studies, each task paradigm is optimized to provide adequate statistical power for single subject mapping, and to be amenable for young children. Additionally, structural MRI studies will allow for in depth tracking of structural changes, including changes in gray-white matter ratios and the integrity of white matter tracts throughout the brain. Blood samples for genetic analysis will be collected. One hundred children with classic Williams syndrome deletions, those with smaller deletions, and those with duplications, along with 50 of their unaffected siblings, will be studied at the NIH Clinical Center at two-year intervals for repeat neuroimaging studies. Additionally, approximately 115 unrelated, healthy children will also be studied. fMRI tasks will be piloted on fifteen of the latter. We will continue to study the children enrolled in this protocol after they turn 18 in order to determine the developmental trajectory of brain structure and function from childhood through adulthood. Additionally, fifty adults with classic Williams syndrome deletions, those with smaller deletions, and those with duplications will be studied at the NIH Clinical Center at two-year intervals for repeat neuroimaging studies in order to establish good adult end-points for our imaging protocol. Studying adults with WS and abnormalities of the WS genetic region with the same tasks and scanner as used for children will allow us to establish an adult WS comparison group against which children can be directly compared and also allow us to better determine the maturation of neural structure and function in WS through adulthood. Typically developing children whom we will continue to study after they turn 18 will serve as the control comparison group for adults with Williams syndrome .

Primary outcome measures include size and integrity of grey and white matter; functional MRI BOLD responses during rest, cognitive and emotion information processing; DTI anisotropy measures of white matter tracts; tissue perfusion (blood flow) measured with arterial spin labeling (ASL); and mcDespot myelin water fraction.

Secondary outcome measures include relationship of neuropsychological assessments and genotyping to the imaging results.

Our prior success in delineating the brain phenotype in adult Williams syndrome patients will provide the crucial context within which to view the emergence and modification of these neural circuit abnormalities from a developmental perspective in children with Williams syndrome and from which to launch translational studies of specific gene effects on brain and behavioral phenotypes.

ELIGIBILITY:
* INCLUSION CRITERIA:

For all participants, the following inclusion criteria will apply:

1. Greater than 5 years old.
2. Able to provide assent if below the age of 18, or consent if 18 years of age or older. Parents will provide consent for participants below the age of 18. For patients who do not have the capacity to provide informed consent, consent may be obtained from a guardian or the holder of the DPA.

Additionally, 7q11.23 CNV participants must have a typical, 7q11.23 CNV or other genetic abnormality in the Williams syndrome critical region of chromosome 7q11.23, and control participants must have normal intelligence.

EXCLUSION CRITERIA:

For all participants who will participate in MRI scanning, the following exclusion criteria will apply:

1. Any chronic or acute medical condition severe enough to interfere with task performance or interpretation of MRI data.
2. Any medication that might interfere with task performance or interpretation of MRI data.
3. Any medical condition that increases risk for MRI (e.g. pacemaker, metallic foreign body in eye or other body part, dental braces).
4. Pregnancy (a urine pregnancy test will be performed prior to all MRI procedures for all females of child-bearing potential.
5. NIMH employees and staff and their immediate family members will be excluded from the study per NIMH policy.

For parents who will undergo blood draws only, they will not be able to participate if they have a condition

that would make collecting blood unsafe.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children with classic WS deletions, those with smaller deletions, and those with duplications of the WS region on chromosome band 7q11.23.
Sampling Method: Probability Sample
Enrollment: 415 (Estimated)
Dates: Start 2011-01-23 (Actual)

PRIMARY OUTCOMES:
fMRI Task Procedures | Ongoing
  fMRI Task Procedures

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Berman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolphs R, Tranel D, Damasio H, Damasio AR. Fear and the human amygdala. J Neurosci. 1995 Sep;15(9):5879-91. doi: 10.1523/JNEUROSCI.15-09-05879.1995. PMID 7666173
- [Background] Ashburner J. A fast diffeomorphic image registration algorithm. Neuroimage. 2007 Oct 15;38(1):95-113. doi: 10.1016/j.neuroimage.2007.07.007. Epub 2007 Jul 18. PMID 17761438
- [Background] Atkinson J, Braddick O, Rose FE, Searcy YM, Wattam-Bell J, Bellugi U. Dorsal-stream motion processing deficits persist into adulthood in Williams syndrome. Neuropsychologia. 2006;44(5):828-33. doi: 10.1016/j.neuropsychologia.2005.08.002. Epub 2005 Sep 15. PMID 16168445
- [Derived] Kippenhan JS, Gregory MD, Nash T, Kohn P, Mervis CB, Eisenberg DP, Garvey MH, Roe K, Morris CA, Kolachana B, Pani AM, Sorcher L, Berman KF. Dorsal visual stream and LIMK1: hemideletion, haplotype, and enduring effects in children with Williams syndrome. J Neurodev Disord. 2023 Aug 26;15(1):29. doi: 10.1186/s11689-023-09493-x. PMID 37633900
- [Derived] Chen G, Nash TA, Cole KM, Kohn PD, Wei SM, Gregory MD, Eisenberg DP, Cox RW, Berman KF, Shane Kippenhan J. Beyond linearity in neuroimaging: Capturing nonlinear relationships with application to longitudinal studies. Neuroimage. 2021 Jun;233:117891. doi: 10.1016/j.neuroimage.2021.117891. Epub 2021 Mar 3. PMID 33667672
- [Derived] Gregory MD, Kolachana B, Yao Y, Nash T, Dickinson D, Eisenberg DP, Mervis CB, Berman KF. A method for determining haploid and triploid genotypes and their association with vascular phenotypes in Williams syndrome and 7q11.23 duplication syndrome. BMC Med Genet. 2018 Apr 4;19(1):53. doi: 10.1186/s12881-018-0563-3. PMID 29614955
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-M-0112.html